CLINICAL TRIAL: NCT03469336
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, VEHICLE AND ACTIVE COMPARATOR-CONTROLLED, PSORIASIS PLAQUE TEST STUDY TO ASSESS SAFETY, TOLERABILITY, AND PSORIATIC SKIN INFILTRATE THICKNESS FOLLOWING REPEATED, TOPICAL DOSES OF PF-06763809 SOLUTION IN SUBJECTS WITH MILD TO MODERATE CHRONIC PLAQUE PSORIASIS
Brief Title: Safety, Tolerability And Efficacy Study Of Topical PF-06763809 In Subjects With Mild To Moderate Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C3561001; 2017-002684-18 (EudraCT Number)
Record Dates: First submitted 2018-03-13; First posted 2018-03-19 (Actual); Results first posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Psoriasis
Keywords: Psoriasis; Topical
MeSH Terms: conditions — Psoriasis | interventions — pf-06763809; calcipotriene; Betamethasone

STUDY DESIGN:
Masking Description: This study is a single arm multi-intervention study. The interventions are masked to participant, investigator, providers and assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- All subjects (Other): All subjects will receive all six interventions/treatments applied to six different treatment fields.
  Interventions: Drug: PF-06763809; Other: Vehicle; Drug: Calcipotriene/calcipotriol; Drug: Betamethasone

INTERVENTIONS:
Drug: PF-06763809 — Three different concentrations will be administered to three different treatment fields: 2.3%, 0.8% and 0.23%
Other: Vehicle — Vehicle matching PF-06763809.
Drug: Calcipotriene/calcipotriol — Calcipotriene/calcipotriol 50 ug/mL solution
Drug: Betamethasone — Betamethasone 1 mg/g solution

SUMMARY:
The study is a randomized, double blinded, vehicle and active comparator controlled, multiple dose study in subjects with chronic plaque psoriasis. The study will have approximately 15 completers. Each subjects will receive three different topical doses of PF 06763809, PF 06763809 vehicle, and two active comparators. These will be applied to six different treatment fields for 18 days. The total duration of participation in the study will be approximately 7 weeks (minimum) to approximately 11 weeks (maximum), including the interval from Screening to the Follow up phone call visit.

ELIGIBILITY:
Inclusion Criteria:

* Psoriasis vulgaris in a chronic stable phase and with a plaque area of mild to moderate severity sufficient for six treatment fields located in up to three plaque areas
* Target lesion(s) should be on the trunk or extremities (excluding palms/soles).

Exclusion Criteria:

* History of skin sensitivity to topical prescription or non prescription products such as creams, lotions and cosmetics
* Psoriasis guttata, psoriasis punctata, psoriasis erythrodermatica, and pustular psoriasis
* Treatment with any biologics within 3 months prior to Day 1 of the study and during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Germany (2):
  - Rothaar Studien GmbH, Berlin
  - bioskin GmbH, Hamburg

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Berstein G, Zhang Y, Berger Z, Kieras E, Li G, Samuel A, Yeoh T, Dowty H, Beaumont K, Wigger-Alberti W, von Mackensen Y, Kroencke U, Hamscho R, Garcet S, Krueger JG, Banfield C, Oemar B. A phase I, randomized, double-blind study to assess the safety, tolerability and efficacy of the topical RORC2 inverse agonist PF-06763809 in participants with mild-to-moderate plaque psoriasis. Clin Exp Dermatol. 2021 Jan;46(1):122-129. doi: 10.1111/ced.14412. Epub 2020 Sep 14. PMID 32767679
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3561001

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 26 participants screened for entry into the study, 4 participants failed at Screening and 4 participants were eligible at Screening but were not randomized in the study, and the remaining 18 participants were assigned to the study treatment.
Groups:
- PF-06763809+Vehicle+Calcipotriene+Betamethasone: All participants with at least 6 test fields received blinded topical doses (2.3%, 0.8% and 0.23%) of PF-06763809, PF-06763809 vehicle, Calcipotriene (50 g/mL) and betamethasone 1 mg/g solution at the six test fields respectively. The dosing volume for all study treatments was 180 µL (164 µL/cm^2), applied topically once daily to 1.1 cm^2 skin surface area of each test field during an 18-day treatment period.
Period: Overall Study
Arm/Group | PF-06763809+Vehicle+Calcipotriene+Betamethasone
Started | 18
Completed | 17
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | PF-06763809+Vehicle+Calcipotriene+Betamethasone
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants] — Age Categorical
  Participants
    <=18 years | 0
    Between 18 and 65 years | 15
    >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Psoriatic Skin Infiltrate Thickness
Description: Baseline was defined to be the measurement on Day 1. MMRM analysis of changes in psoriatic skin in psoriatic skin infiltrate thickness/echo poor band (EPB) in response to PF-06763809 2.3%, 0.8% and 0.23% applied topically for 18 consecutive days as compared to the vehicle control. Number of participants analyzed signifies number of participants who were evaluable for this outcome measure. Number analyzed refers to number of participants evaluable for specified rows of categories.
Time Frame: Baseline, Days 7, 13 and 19
Population: Analysis population included all participants who had at least one application of the investigational products and had at least one post-baseline assessment of the primary efficacy variable, were included in the Full Analysis Set (FAS).
Measure: Geometric Mean (Standard Error); unit: micrometer (μm)
Groups:
- A: PF-06763809 2.3% Solution: Participants were exposed to 2.3% PF-06763809 solution once daily during an 18-day treatment period. Daily dosage: approximately 4.1 mg PF-06763809. Total dosage: approximately 75 mg PF-06763809
- B: PF-06763809 0.8% Solution: Participants were exposed to 0.8% PF-06763809 solution once daily during an 18-day treatment period. Daily dosage: approximately 1.4 mg PF-06763809. Total dosage: approximately 26 mg PF-06763809
- C: PF-06763809 0.23% Solution: Participants were exposed to 0.23% PF-06763809 solution once daily during an 18-day treatment period. Daily dosage: approximately 0.41 mg PF-06763809. Total dosage: approximately 7.5 mg PF-06763809.
- D: PF-06763809 Vehicle: Participants were exposed to active ingredient-free vehicle to PF-06763809 treatments once daily during an 18-day treatment period.
Arm/Group | A: PF-06763809 2.3% Solution | B: PF-06763809 0.8% Solution | C: PF-06763809 0.23% Solution | D: PF-06763809 Vehicle
Number analyzed (Participants) | 18 | 18 | 18 | 18
micrometer (μm)
  Day 7 | 0.89 (0.073) | 0.92 (0.073) | 0.97 (0.073) | 0.93 (0.073)
  Day 13: number analyzed (Participants) | 17 | 17 | 18 | 17
  Day 13 | 0.74 (0.458) | 0.76 (0.458) | 0.87 (0.458) | 0.80 (0.458)
  Day 19: number analyzed (Participants) | 17 | 17 | 18 | 17
  Day 19 | 0.71 (0.526) | 0.70 (0.526) | 0.80 (0.526) | 0.70 (0.526)
Statistical Analysis 1: Comparison: A: PF-06763809 2.3% Solution vs D: PF-06763809 Vehicle; The efficacy assessment of PF-06763809 was performed for the change from baseline in log of the psoriatic skin infiltrate thickness/EPB on Day 19 using a longitudinal analysis of covariance model, with treatment, visit, treatment by visit interaction as main effects and the log of the psoriatic skin infiltrate thickness/EPB at baseline as covariate; Test type: Other — Ratio; p = 0.9883, Mixed Models Analysis; Mean Ratio (Test/Reference) = 1.0109, 95% CI 2-sided [0.2364 to 4.3226], Standard Error of Mean 0.732
Statistical Analysis 2: Comparison: B: PF-06763809 0.8% Solution vs D: PF-06763809 Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Other — Ratio; p = 0.9977, Mixed Models Analysis; Mean Ratio (Test/Reference) = 0.9979, 95% CI 2-sided [0.2334 to 4.2671], Standard Error of Mean 0.732
Statistical Analysis 3: Comparison: C: PF-06763809 0.23% Solution vs D: PF-06763809 Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Other — Ratio; p = 0.8600, Mixed Models Analysis; Mean Ratio (Test/Reference) = 1.1382, 95% CI 2-sided [0.2662 to 4.8670], Standard Error of Mean 0.732

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs)
Description: Baseline was defined to be the measurement on Day 1. An AE was any untoward medical occurrence in a clinical investigation patient administered a product or medical device. Treatment-emergent AEs were those with initial onset or increasing in severity after the first dose of investigational product.
Time Frame: Day 1 to Day 49
Population: Analysis population included all participants who received at least one application of the investigational products and had at least one post-baseline efficacy assessment value.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06763809+Vehicle+Calcipotriene+Betamethasone
Number analyzed (Participants) | 18
Participants | 6

3. Primary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: Baseline was defined to be the measurement on Day 1. The safety laboratory tests including Hematology, Clinical Chemistry and Urinalysis were performed. Hematology evaluation included: hemoglobin (HGB) (gram per decilitre=g/dL), hematocrit, erythrocytes (Ery.), Ery. Mean Corpuscular Volume, Ery. Mean Corpuscular Hemoglobin, Ery. Mean Corpuscular HGB Concentration (picograms per cell=pg/cell), platelets, leukocytes, lymphocytes, and neutrophils. Clinical chemistry evaluation included: bilirubin, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, protein, albumin, urea nitrogen, urea, creatinine, urate, sodium, potassium, chloride, calcium, bicarbonate, creatine kinase, and glucose. Urinalysis evaluation included: pH, urine glucose, ketones, urine protein, urine hemoglobin, urobilinogen, urine bilirubin, nitrite, and leukocyte esterase. LLN=lower limit of normal, ULN=upper limit of normal.
Time Frame: Day 1 to Day 49
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06763809+Vehicle+Calcipotriene+Betamethasone
Number analyzed (Participants) | 18
Participants
  Hemoglobin (HGB) (g/dL) <0.8xLLN | 0
  Hematocrit (%) <0.8xLLN | 0
  Erythrocytes (10^6/mm^3) <0.8xLLN | 0
  Ery. Mean Corpuscular Volume (μm^3) <0.9xLLN | 0
  Ery. Mean Corpuscular Volume (μm^3) >1.1xULN | 1
  Ery. Mean Corpuscular HGB (pg/cell) <0.9xLLN | 0
  Ery. Mean Corpuscular HGB (pg/cell) >1.1xULN | 0
  Ery. Mean Corpuscular HGB Conc. (g/dL) <0.9xLLN | 1
  Ery. Mean Corpuscular HGB Conc. (g/dL) >1.1xULN | 0
  Platelets (10^3/mm^3) <0.5xLLN | 0
  Platelets (10^3/mm^3) >1.75xULN | 0
  Leukocytes (10^3/mm^3) <0.6xLLN | 0
  Leukocytes (10^3/mm^3) >1.5xULN | 0
  Lymphocytes (10^3/mm^3) <0.8xLLN | 2
  Lymphocytes (10^3/mm^3) >1.2xULN | 0
  Neutrophils (10^3/mm^3) <0.8xLLN | 0
  Neutrophils (10^3/mm^3) >1.2xULN | 0
  Basophils (10^3/mm^3) >1.2xULN | 0
  Eosinophils (10^3/mm^3) >1.2xULN | 0
  Monocytes (10^3/mm^3) >1.2xULN | 1
  Bilirubin (mg/dL) >1.5xULN | 0
  Aspartate Aminotransferase (U/L) >3.0xULN | 0
  Alanine Aminotransferase (U/L) >3.0xULN | 0
  Alkaline Phosphatase (U/L) >3.0xULN | 0
  Protein (g/dL) <0.8xLLN | 0
  Protein (g/dL) >1.2xULN | 0
  Albumin (g/dL) <0.8x LLN | 0
  Albumin (g/dL) >1.2xULN | 0
  Urea Nitrogen (mg/dL) >1.3xULN | 0
  Urea (mmol/L) >1.3xULN | 0
  Creatinine (mg/dL) >1.3xULN | 0
  Urate (mg/dL) >1.2xULN | 0
  Sodium (mEq/L) <0.95xLLN | 0
  Sodium (mEq/L) >1.05xULN | 0
  Potassium (mEq/L) <0.9x LLN | 0
  Potassium (mEq/L) >1.1xULN | 0
  Chloride (mEq/L) <0.9xLLN | 0
  Chloride (mEq/L) >1.1xULN | 0
  Calcium (mg/dL) <0.9x LLN | 0
  Calcium (mg/dL) >1.1xULN | 0
  Bicarbonate (mEq/L) <0.9x LLN | 0
  Bicarbonate (mEq/L) >1.1xULN | 0
  Glucose (mg/dL) <0.6xLLN | 0
  Glucose (mg/dL) >1.5xULN | 0
  pH (Scalar) <4.5 | 0
  pH (Scalar) >8 | 0
  URINE Glucose (Scalar) >=1 | 0
  Ketones (Scalar) >=1 | 0
  URINE Protein (Scalar) >=1 | 0
  URINE Hemoglobin (Scalar) >=1 | 0
  Urobilinogen (Scalar) >=1 | 0
  URINE Bilirubin (Scalar) >=1 | 0
  Nitrite (Scalar) >=1 | 0
  Leukocyte Esterase (Scalar) >=1 | 0

4. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting Pre-specified Criteria
Description: Baseline was defined to be the measurement on Day 1. ECG categorical summarization criteria: 1) PR interval (Value>=300 milliseconds [msec], %Change [Chg]>=25/50%); 2) QRS interval (Value>=140 msec, >=50% change from baseline; 2) PR interval (the interval between the start of the P wave and the start of the QRS complex, corresponding to the time between the onset of the atrial depolarization and onset of ventricular depolarization): >=300 msec, >=25% change when baseline is > 200 msec or >=50% change when baseline is less than or equal to (<=) 200 msec; 3) QT interval (time from ECG Q wave to the end of the T wave corresponding to electrical systole): absolute value of >=500 msec; 4) QTc interval (QT corrected for heart rate): absolute value of 450 to <480 msec, 480 to <500 msec, >=500 msec; a change from baseline of 30 to <60 msec or >=60 msec. The corrected QT interval by Fredericia=QTcF Interval.
Time Frame: Day 1 to Day 49
Population: Analysis population included all participants who received at least one application of the investigational products and had at least one post-baseline efficacy assessment value. All scheduled ECGs were performed after the participant had rested quietly for 10 minutes in a supine position.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06763809+Vehicle+Calcipotriene+Betamethasone
Number analyzed (Participants) | 18
Participants
  Value>=300 msec (PR Interval) | 0
  %Change (Chg)>=25/50% (PR Interval) | 0
  Value>=140 msec (QRS Interval) | 0
  %Chg>=50% (QRS Interval) | 0
  Value>=500 msec (QT Interval) | 0
  450<=Value<480 msec (QTc Interval) | 2
  480<=Value<500 msec (QTc Interval) | 0
  Value>=500 msec (QTc Interval) | 0
  30<=Chg<60 msec (QTc Interval) | 2
  Chg>=60 msec (QTc Interval) | 1
  450<=Value<480 msec (QTcF Interval) | 0
  480<=Value<500 msec (QTcF Interval) | 0
  Value>=500 msec (QTcF Interval) | 0
  30<=Chg<60 msec (QTcF Interval) | 0
  Chg>=60 msec (QTcF Interval) | 0

5. Primary Outcome: Number of Participants With Post-Baseline Vital Signs Data Meeting Categorical Summarization Criteria
Description: Baseline was defined to be the measurement on Day 1. Vital Signs including diastolic blood pressure (DBP), pulse rate, and systolic blood pressure (SBP) were measured.
Time Frame: Day 1 to Day 49
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06763809+Vehicle+Calcipotriene+Betamethasone
Number analyzed (Participants) | 18
Participants
  DBP Value <50 mmHg | 0
  DBP Chg >= 20 mmHg increase | 0
  DBP Chg >= 20 mmHg decrease | 0
  Pulse Rate Value <40 beats per minute (bpm) | 0
  Pulse Rate Value >120 bpm | 0
  SBP Value <90 mmHg | 0
  SBP Chg >= 30 mmHg increase | 0
  SBP Chg >= 30 mmHg decrease | 0

6. Secondary Outcome: Area Under the Curve of the Psoriatic Skin Infiltrate Thickness
Description: Baseline was defined to be the measurement on Day 1. To evaluate the Area Under the Curve (AUC) of psoriatic skin infiltrate thickness/EPB for PF 06763809 compared to vehicle by mixed model analysis. The AUC of the psoriatic skin infiltrate thickness/EPB from Day 1 to Day 19 was determined using the linear trapezoidal rule. The log AUC was performed by the natural logarithm of the AUC of the psoriatic skin infiltrate thickness/EPB. Number of participants analyzed signifies number of participants who were evaluable for this outcome measure. Number analyzed refers to number of participants evaluable for specified rows of categories.
Time Frame: Day 1 to Day 19
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: nanograms*hour per milliliter (ng*h/mL)
Arm/Group | A: PF-06763809 2.3% Solution | B: PF-06763809 0.8% Solution | C: PF-06763809 0.23% Solution | D: PF-06763809 Vehicle
Number analyzed (Participants) | 18 | 18 | 18 | 18
nanograms*hour per milliliter (ng*h/mL) | 6191.52 (0.124) | 5996.26 (0.115) | 6921.58 (0.107) | 6204.82 (0.094)
Statistical Analysis 1: Comparison: A: PF-06763809 2.3% Solution vs D: PF-06763809 Vehicle; To evaluate the AUC of psoriatic skin infiltrate thickness/EPB for PF-06763809 compared to vehicle; Test type: Other — Ratio; p = 0.9763, Mixed Models Analysis; Mean Ratio (Test/Reference) = 0.9979, 95% CI 2-sided [0.8588 to 1.1594], Standard Error of Mean 0.071
Statistical Analysis 2: Comparison: B: PF-06763809 0.8% Solution vs D: PF-06763809 Vehicle; To evaluate the AUC of psoriatic skin infiltrate thickness/EPB for PF-06763809 compared to vehicle; Test type: Other — Ratio; p = 0.5081, Mixed Models Analysis; Mean Ratio (Test/Reference) = 0.9664, 95% CI 2-sided [0.8686 to 1.0752], Standard Error of Mean 0.051
Statistical Analysis 3: Comparison: C: PF-06763809 0.23% Solution vs D: PF-06763809 Vehicle; To evaluate the AUC of psoriatic skin infiltrate thickness/EPB for PF-06763809 compared to vehicle; Test type: Other — Ratio; p = 0.0249, Mixed Models Analysis; Mean Ratio (Test/Reference) = 1.1155, 95% CI 2-sided [1.0157 to 1.2252], Standard Error of Mean 0.044

7. Secondary Outcome: Change From Baseline in Skin Infiltrate Thickness in Response to PF-06763809 Compared to Calcipotriene/Calcipotriol Solution.
Description: The effect of PF-06763809 compared to calcipotriene/calcipotriol solution in the change of psoriatic skin infiltrate thickness/EPB both within and following 18 days of treatment. Baseline was defined to be the measurement on Day 1. Number of participants analyzed signifies number of participants who were evaluable for this outcome measure. Number analyzed refers to number of participants evaluable for specified rows of categories.
Time Frame: Baseline, Days 7, 13 and 19
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: μm
Groups:
- E: Calcipotriene/Calcipotriol Solution: Participants were exposed to Calcipotriene/ calcipotriol (50 g/mL) once daily during an 18-day treatment period. Daily dosage of calcipotriol: approximately 0.01 mg. Total dosage: approximately 0.18 mg.
Arm/Group | A: PF-06763809 2.3% Solution | B: PF-06763809 0.8% Solution | C: PF-06763809 0.23% Solution | E: Calcipotriene/Calcipotriol Solution
Number analyzed (Participants) | 18 | 18 | 18 | 18
μm
  Day 7 | 0.89 (0.073) | 0.92 (0.073) | 0.97 (0.073) | 0.77 (0.073)
  Day 13: number analyzed (Participants) | 17 | 17 | 18 | 17
  Day 13 | 0.74 (0.458) | 0.76 (0.458) | 0.87 (0.458) | 0.86 (0.458)
  Day 19: number analyzed (Participants) | 17 | 17 | 18 | 17
  Day 19 | 0.71 (0.526) | 0.70 (0.526) | 0.80 (0.526) | 0.90 (0.526)
Statistical Analysis 1: Comparison: A: PF-06763809 2.3% Solution vs E: Calcipotriene/Calcipotriol Solution; The effect of PF-06763809 compared to calcipotriene/calcipotriol solution in the change of psoriatic skin infiltrate thickness/EPB on Day 19; Test type: Other — Ratio; p = 0.7540, Mixed Models Analysis; Mean Ratio (Test/Reference) = 0.7946, 95% CI 2-sided [0.1858 to 3.3977], Standard Error of Mean 0.732
Statistical Analysis 2: Comparison: B: PF-06763809 0.8% Solution vs E: Calcipotriene/Calcipotriol Solution; [analysis description as in outcome 7, analysis 1]; Test type: Other — Ratio; p = 0.7407, Mixed Models Analysis; Mean Ratio (Test/Reference) = 0.7844, 95% CI 2-sided [0.1834 to 3.3540], Standard Error of Mean 0.732
Statistical Analysis 3: Comparison: C: PF-06763809 0.23% Solution vs E: Calcipotriene/Calcipotriol Solution; [analysis description as in outcome 7, analysis 1]; Test type: Other — Ratio; p = 0.8793, Mixed Models Analysis; Mean Ratio (Test/Reference) = 0.8946, 95% CI 2-sided [0.2092 to 3.8256], Standard Error of Mean 0.732

8. Secondary Outcome: Change From Baseline in Skin Infiltrate Thickness in Response to PF-06763809 Compared to Betamethasone Solution.
Description: The effect of PF-06763809 compared to betamethasone solution in the change of psoriatic skin infiltrate thickness/EPB both within and following 18 days of treatment. Baseline was defined to be the measurement on Day 1. Number of participants analyzed signifies number of participants who were evaluable for this outcome measure. Number analyzed refers to number of participants evaluable for specified rows of categories.
Time Frame: Baseline, Days 7, 13 and 19
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: μm
Groups:
- F: Betamethasone Solution.: Participants were exposed to Betamethasone (1 mg/g) once daily during an 18-day treatment period. Daily dosage of approximately 0.18 mg. Total dosage: approximately 3.2 mg.
Arm/Group | A: PF-06763809 2.3% Solution | B: PF-06763809 0.8% Solution | C: PF-06763809 0.23% Solution | F: Betamethasone Solution.
Number analyzed (Participants) | 18 | 18 | 18 | 18
μm
  Day 7 | 0.89 (0.073) | 0.92 (0.073) | 0.97 (0.073) | 0.43 (0.073)
  Day 13: number analyzed (Participants) | 17 | 17 | 18 | 17
  Day 13 | 0.74 (0.458) | 0.76 (0.458) | 0.87 (0.458) | 0.03 (0.458)
  Day 19: number analyzed (Participants) | 17 | 17 | 18 | 17
  Day 19 | 0.71 (0.526) | 0.70 (0.526) | 0.80 (0.526) | 0.01 (0.526)
Statistical Analysis 1: Comparison: A: PF-06763809 2.3% Solution vs F: Betamethasone Solution; The effect of PF-06763809 compared to betamethasone solution in the change of psoriatic skin infiltrate thickness/EPB on Day 19; Test type: Other — Ratio; p < 0.0001, Mixed Models Analysis; Mean Ratio (Test/Reference) = 1.081321, 95% CI 2-sided [0.25287 to 4.623941], Standard Error of Mean 0.732
Statistical Analysis 2: Comparison: B: PF-06763809 0.8% Solution vs F: Betamethasone Solution; [analysis description as in outcome 8, analysis 1]; Test type: Other — Ratio; p < 0.0001, Mixed Models Analysis; Mean Ratio (Test/Reference) = 1.067453, 95% CI 2-sided [0.249631 to 4.564555], Standard Error of Mean 0.732
Statistical Analysis 3: Comparison: C: PF-06763809 0.23% Solution vs F: Betamethasone Solution; [analysis description as in outcome 8, analysis 1]; Test type: Other — Ratio; p < 0.0001, Mixed Models Analysis; Mean Ratio (Test/Reference) = 1.217483, 95% CI 2-sided [0.284708 to 5.206258], Standard Error of Mean 0.732

ADVERSE EVENTS:
Time Frame: Day 1 to Day 49
Description: All Participants with a treatment area sufficient for 6 treatment fields received topical doses (2.3%, 0.8% and 0.23%) of PF-06763809, vehicle, Calcipotriene (50 g/mL) and betamethasone 1 mg/g solution at 6 test areas, respectively. Therefore, although treatment-emergent skin-related AEs could tell which treatment caused the AE, other treatment-emergent AEs not related to a specific treatment area could not be assigned to a treatment and were reported for the entire participant population.
Arm/Group | PF-06763809+Vehicle+Calcipotriene+Betamethasone
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 6/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-06763809+Vehicle+Calcipotriene+Betamethasone (N=18)
Blepharitis (Eye disorders) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) — One (1) TEAE of acute exacerbation of Psoriasis (severe in severity) was reported independent of treatment field and was considered not treatment-related by the investigator.
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4 (4) — Four treatment-emergent skin-related AEs of Dermatitis contact were all reported on the Calcipotriene (50 g/mL) solution treated fields.
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) — One (1) treatment-emergent skin related TEAE of Pruritus was reported on PF-06763809 vehicle treated field.
Nasopharyngitis (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-04-03): https://cdn.clinicaltrials.gov/large-docs/36/NCT03469336/SAP_000.pdf
  • Study Protocol (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/36/NCT03469336/Prot_001.pdf